CLINICAL TRIAL: NCT05439434
Title: Turkish Reliability and Validity of The Fear of Pain Questionnaire for Children Short Form (FOPQC-SF) in Children/Adolescents With Juvenile Idiopathic Arthritis
Brief Title: Turkish Reliability and Validity of FOPQC-SF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Elif Gur Kabul, Pirincipal Investigator, Pamukkale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FOPQC-SF
Record Dates: First submitted 2022-06-26; First posted 2022-06-30 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Fear; Pain; Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Pain; Arthritis, Juvenile

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention group (Experimental)
  Interventions: Other: Fear of Pain Questionnaire for Children Short Form

INTERVENTIONS:
Other: Fear of Pain Questionnaire for Children Short Form — administering the questionnaire twice, one week apart.

SUMMARY:
The aim of this study is to question the Turkish validity and reliability of the "The Fear of Pain Questionnaire for Children Short Form (FOPQC-SF)" scale. Children/adolescents between the ages of 7-18 and diagnosed with Juvenile Idiopathic Arthritis followed by the Pediatric Rheumatology Clinic will be included in the study. The sample size of this study was determined as at least 50. To assess the validity of the FOPQC-SF scale, participants will be administered the Pediatric Quality of Life Inventory (PedsQL) 3.0 Arthritis Module, the Childhood Health Assessment Questionnaire (CHAQ), and the Juvenile Arthritis Disease Activity Score.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with JIA according to the ILAR classification
* 7-18 years old
* Agree to participate in the study

Exclusion Criteria:

* Psychiatric illness that may affect cooperation,
* Those with heart failure and lung pathology at a level that will affect their daily life activities

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Fear of Pain Questionnaire for Children Short Form | 10 minutes
  It consists of 10 items in total. All items are scored between O-4. Higher scores indicate higher levels of pain-related fear and avoidance.

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory (PedsQL) 3.0 Arthritis Module | 15 minutes
  Total score ranging from 0-100. High scores mean high quality of life.
Juvenile Arthritis Disease Activity Score | 10 minutes
  Total JADAS score ranging from 0-57. Higher score indicates more disease activity.
Childhood Health Assessment Questionnaire | 15 minutes
  It consists of 8 subtests and 30 questions. It is scored between 0-3. A higher score indicates more disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Pamukkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No